CLINICAL TRIAL: NCT01677078
Title: Assessment of the Neuronavigation System Coupled With Repetitive Transcranial Magnetic Stimulation. A Randomized Double Blind Study
Brief Title: Coupling Repetitive Transcranial Magnetic Stimulation With a Neuronavigation System in Treatment Resistant Depression
Acronym: TMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-A01272-39
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Treatment Resistant Depression
Keywords: Major depressive disorder; rTMS; Neuronavigation
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuronavigation system (Experimental): 10 sessions of rTMS coupled with a neuronavigation system
  Description of 1 session of the rTMS protocol :
  * Frequency: 20Hz
  * Intensity: 110% of motor threshold
  * 80 train of 2 seconds duration
  * 10 seconds between two trains
  * 3200 pulses
  Devices :
  * rTMS: System Mag Pro (Magventure, Denmark)
  * Neuronavigation system: Syneika One (Syneika, France)
  Interventions: Device: Neuronavigation system
- Standard localisation method (Sham Comparator): 10 sessions of rTMS with manual localisation of the DLPFC using the standard localisation method (i.e. the '5-cm method')
  Description of 1 session of the rTMS protocol :
  * Frequency: 20Hz
  * Intensity: 110% of motor threshold
  * 80 train of 2 seconds duration
  * 10 seconds between two trains
  * 3200 pulses
  Devices :
  - rTMS: System Mag Pro (Magventure, Denmark)
  Interventions: Device: Standard localisation method

INTERVENTIONS:
Device: Neuronavigation system — Neuronavigation
  Other Names: Syneika One (Syneika, France)
  Arms: Neuronavigation system
Device: Standard localisation method — Manual localisation of the DLPFC using the standard localisation method (i.e. the '5-cm method')
  Arms: Standard localisation method

SUMMARY:
Repetitive Transcranial Magnetic Stimulation (rTMS) is a non invasive technique which was shown to be effective in the treatment of major depression.

The dorsolateral prefrontal cortex (DLPFC) is the anatomic target in rTMS studies and the standard (manual) '5-cm method' for positioning the coil over DLPFC is the reference. Nevertheless, it has been criticized due to poor targeting accuracies attributed to inter-subject variability.

Such an inaccuracy could have any therapeutic consequences as a decrease in rTMS efficacy.

Preliminary findings suggest that a more reproductible and accurate method, based upon a neuronavigation system could allow for a better efficacy. This finding has to be replicated with sound methodology.

Investigator's objective is to compare efficacy on mood of coil positioning based upon a neuronavigation device versus coil positioning based upon the standard method.

DETAILED DESCRIPTION:
Background :

Repetitive Transcranial Magnetic Stimulation (rTMS) is a new tool for major depressive disorder.

rTMS is a non invasive technique allowing for a localized stimulation of cerebral tissue cortex. rTMS uses electromagnetic induction to induce weak electric currents using a rapidly changing magnetic field; this can modify activity in specific or general parts of the brain.

Meta-analyses have stated that rTMS appeared to be effective in the treatment of major depression despite any limits concerning sample sizes and methodological concerns.

Studies have shown that this technique potentiates antidepressants treatment in combination therapy.

It has received FDA approval for the management of major depressive disorder. Stimulation parameters are numerous (frequency, intensity, number of pulses) and their effects are increasingly better understood in order to predict a better balance between efficacy and tolerability.

The dorsolateral prefrontal cortex (DLPFC) is the target in repetitive transcranial magnetic stimulation and the standard (manual) '5-cm method' for positioning the transcranial magnetic stimulation coil over DLPFC is the reference. It has been criticized due to poor targeting accuracies attributed to inter-subject variability.

Such an inaccuracy could have consequences as a decrease in rTMS efficacy. Any preliminary findings suggest that a more reproductible and accurate method, based upon a neuronavigation system could allow for a better efficacy. This finding has to be replicated with sound methodology.

Objectives:

To compare efficacy on mood of coil positioning based upon a neuronavigation device versus coil positioning based upon the standard method.

Investigators hypothesized that an accurate localization and stimulation of DLPFC using neuronavigation would be more effective than the less accurate standard method.

A secondary objective is to compare the efficacy on patient's self perception, on psychomotor symptoms and the tolerability of the two methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients giving their consent;
* Right handed;
* Age > 18 and < 65;
* With a DSM-IV diagnosis of MDD, single episode or recurrent;
* With an antidepressant treatment unchanged in the 3 last weeks;
* With an MADRS score ≥ 21;
* Benzodiazepine treatments have to be avoided;

Exclusion Criteria:

* Major depressive episode with psychotic characteristics;
* A lifetime of the following axis 1 diagnoses: schizophrenia or substance use disorder (alcohol or other substance);
* Stade 5 of Thase and Rush classification ;
* Involuntary hospitalizations;
* Patients under guardianship;
* Outpatients in case of an increased risk of suicide as assessed by a MADRS item 10 > 3;
* Contraindication for MRI or rTMS: a personal history of a seizure disorder, presence of neurologic or neurosurgical disorder, presence of ferromagnetic material (including intraocular) or metallic medical devices (pacemakers);
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2013-01-21 (Actual); Primary Completion 2017-03-25 (Actual); Study Completion 2017-03-25 (Actual)

PRIMARY OUTCOMES:
Response | Day 44
  Response defined as at least 50% reduction in the MADRS score.

SECONDARY OUTCOMES:
Response | Day 14
  Response is defined as at least 50% reduction in the MADRS score.
Remission | Day 14 Day 44
  Remission is defined as a MADRS score ≤ 8.
MADRS | Day 0, day 14 and day 44
  Description: It is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders.
BDI | Day 0 Day 14 Day 14
  It is a multiple-choice self-report inventory and one of the most widely used instruments for measuring the severity of depression.
ERD | Day 0 Day 14 day 44
  It is a 14-item questionnaire which psychiatrists use to measure the intensity of motor retardation.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Millet, MD PhD, Principal Investigator — CHU Rennes; Jean Michel Reymann, PhD, Study Chair — CHU Rennes
Locations (5):
- France (5):
  - Centre Santé Mentale Angevin CESAME, Angers
  - CHU de Brest, Brest
  - Etablissement Public de Santé Mentale, Quimperlé
  - CHGR, Rennes
  - EPSM Morbihan, Saint-Avé

REFERENCES:
- [Derived] Millet B, Harika-Germaneau G, Maatoug R, Naudet F, Reymann JM, Turmel V, Batail JM, Soulabaille J, Jaafari N, Drapier D. Repetitive Transcranial Magnetic Stimulation targeted with MRI based neuro-navigation in major depressive episode: a double-blind, multicenter randomized controlled trial. PLoS One. 2025 May 27;20(5):e0317597. doi: 10.1371/journal.pone.0317597. eCollection 2025. PMID 40424301